CLINICAL TRIAL: NCT05277467
Title: Urinary Incontinence in Elderly Patients and Its Impact on Caregiver Burden: An Overlooked and Underestimated Topic
Brief Title: Elderly Urinary Incontinence Caregiver Burden
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Other Study IDs: 22
Record Dates: First submitted 2022-02-01; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Caregiver Burden; Urinary Incontinence
Keywords: urinary incontinence; elderly patient; family member; caregiver; caregiver burden
MeSH Terms: conditions — Caregiver Burden; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of this study is to evaluate the severity of urinary incontinence (UI) in elderly patients and its impact on the burden of care in their family caregivers.

DETAILED DESCRIPTION:
The objective was to evaluate the severity of urinary incontinence (UI) in elderly patients and its impact on the burden of care in their family caregivers.

The study is a descriptive, cross-sectional and relationship-seeking type of research. It was conducted prospectively with 80 elderly(≥65 years of age) patients with UI and their family caregivers who applied to the urology clinic between June and December 2021. The data was collected using the "Socio-Demographic Characteristics Data Collection Form". UI was assessed by "International Consultation on Incontinence Questionnaire Short Form(ICIQ-UI-SF)" and caregiver burden by means of Zarit Burden Scale(ZBI) form.

ELIGIBILITY:
Inclusion Criteria:

* The primary caregiver family member (mother, father, spouse, sibling, child), appropriate cognitive and mental health to respond to the applied forms, constant patient care
* The patient's being 65 years and older and diagnosed with urinary incontinence.

Exclusion Criteria:

* The family member who did not volunteer to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study was conducted prospectively with 80 elderly (≥65 years of age) patients with UI and their family caregivers who applied to the urology clinic of a state hospital between June and December 2021 and who have agreed to the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form | This form was applied to the patients immediately after the patient examination at the urology clinic.
  It is a reliable and useful form developed to examine the effect of UI on quality of life. There are questions on the scale that include evaluating the effect of UI on frequency, amount, causes and burden of care. The scale is of likert type and consists of four dimensions. The first dimension includes the frequency of the UI, the second dimension the amount of the UI, the third dimension the impact of the UI on daily life, and the fourth dimension the situations that cause the UI. The maximum score that can be obtained from the scale is 21, and 8 points and above define the UI that causes discomfort.
Zarit Burden Interview | This form was applied to the patients immediately after the patient examination at the urology clinic.
  The caregiving burden scale was used to evaluate the difficulty of providing care experienced by caregivers. 0-20 points from the scale indicate "never a burden of care'', 21-40 points indicate "burden of care rarely'', 41-60 points indicate "burden of care quite frequently'' and 61-88 points indicate "burden of care nearly always''.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay BEKTAS AKPINAR, PhD, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eifert EK, Adams R, Dudley W, Perko M. Family caregiver identity: A literature review. American Journal of Health Education. 2015;46(6):357-67.
- [Background] D'Ancona C, Haylen B, Oelke M, Abranches-Monteiro L, Arnold E, Goldman H, Hamid R, Homma Y, Marcelissen T, Rademakers K, Schizas A, Singla A, Soto I, Tse V, de Wachter S, Herschorn S; Standardisation Steering Committee ICS and the ICS Working Group on Terminology for Male Lower Urinary Tract & Pelvic Floor Symptoms and Dysfunction. The International Continence Society (ICS) report on the terminology for adult male lower urinary tract and pelvic floor symptoms and dysfunction. Neurourol Urodyn. 2019 Feb;38(2):433-477. doi: 10.1002/nau.23897. Epub 2019 Jan 25. PMID 30681183
- [Result] Talley KMC, Davis NJ, Peden-McAlpine C, Martin CL, Weinfurter EV, Wyman JF. Navigating through incontinence: A qualitative systematic review and meta-aggregation of the experiences of family caregivers. Int J Nurs Stud. 2021 Nov;123:104062. doi: 10.1016/j.ijnurstu.2021.104062. Epub 2021 Aug 13. PMID 34461378
- [Result] Yang E, Lisha NE, Walter L, Obedin-Maliver J, Huang AJ. Urinary Incontinence in a National Cohort of Older Women: Implications for Caregiving and Care Dependence. J Womens Health (Larchmt). 2018 Sep;27(9):1097-1103. doi: 10.1089/jwh.2017.6891. Epub 2018 Jun 14. PMID 29902123
- [Result] Yenisehir S, Citak Karakaya I, Karakaya MG. Knowledge and practice of nursing home caregivers about urinary incontinence. Eur Geriatr Med. 2019 Feb;10(1):99-105. doi: 10.1007/s41999-018-0129-0. Epub 2018 Nov 13. PMID 32720273
- [Result] Di Rosa M, Lamura G. The impact of incontinence management on informal caregivers' quality of life. Aging Clin Exp Res. 2016 Feb;28(1):89-97. doi: 10.1007/s40520-015-0367-7. Epub 2015 May 10. PMID 25957737
- [Result] Davis NJ, Parker VG, Lanham J, Love CR, Christy MR, Poetzschke E, Wyman JF. Burdens and Educational Needs of Informal Caregivers of Older Adults With Urinary Incontinence: An Internet-Based Study. Rehabil Nurs. 2021 May-Jun 01;46(3):172-178. doi: 10.1097/rnj.0000000000000317. PMID 33591086